CLINICAL TRIAL: NCT06345599
Title: Phase I+Phase II Clinical Study of PRaG Therapy in Combination With Chemotherapy (AG Regimen) for Neoadjuvant Treatment of Locally Advanced Pancreatic Ductal Adenocarcinoma (PDAC) (NeoPRAG Study)
Brief Title: PRaG Therapy in Combination With Locally Advanced Pancreatic Ductal Adenocarcinoma (PDAC) (NeoPRAG Study)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LK2023100
Record Dates: First submitted 2024-02-01; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Locally Advanced Pancreatic Ductal Adenocarcinoma; Chemotherapy; Neoadjuvant Treatment; PRaG Therapy
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Radiotherapy、Immunotherapy、Chemotherapy
  Interventions: Radiation: Radiotherapy; Drug: Immunotherapy:Granulocyte macrophage-colony stimulating factor(GM-CSF)、Cadumilimab; Drug: Chemotherapy:Albumin-bound paclitaxel、Gemcitabine

INTERVENTIONS:
Radiation: Radiotherapy — This study is a phase I clinical study. The study is divided into phases Ia and Ib. Phase Ia is a dose-escalation experiment, divided into two cohorts based on radiotherapy dose, with 3+3 patients per cohort for a total of 12 patients. The first group undergoes two cycles of radiotherapy: 24Gy:8Gy3f d4-d6. The second group undergoes one cycle of radiotherapy: 40Gy:8Gy5f d3-d7. Phase II consists of 40 patients who choose the radiotherapy dose based on the results of phase I.
Drug: Immunotherapy:Granulocyte macrophage-colony stimulating factor(GM-CSF)、Cadumilimab — GM-CSF treatment: GM-CSF 200μg was started on the day of radiotherapy, and was subcutaneously injected daily for 7 consecutive days; d1-d7 Cadumilimab: use 375mg of cadumilimab within one week after radiotherapy
Drug: Chemotherapy:Albumin-bound paclitaxel、Gemcitabine — Albumin-bound paclitaxel 125mg/m2 d1, d8 Gemcitabine 1000mg/m2 d1, d8 After 3 cycles of neoadjuvant combination treatment with cadumilimab, the patient's surgical status will be evaluated. If surgery is possible, the patient will continue with another 3 cycles of treatment post-operation.

SUMMARY:
The goal of this clinical trial is to learn about Phase I+Phase II Clinical Study of PRaG Therapy in Combination With Chemotherapy (AG Regimen) for Neoadjuvant Treatment of Locally Advanced Pancreatic Ductal Adenocarcinoma (PDAC) (NeoPRAG Study).The main question it aims to answer is to investigate the safety and efficacy of the PRaG treatment modality combined with chemotherapy neoadjuvant therapy for locally advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 ≤ 75 years；no gender limitations
* Histopathologically and/or cytologically confirmed ductal adenocarcinoma of the pancreas, the patient has fresh pathological tissue and the tumour is located in the head and neck or body of the pancreas
* Locally advanced pancreatic cancer, borderline resectable or unresectable, without metastases.
* Life expectancy >= 3 months.
* ECOG score 0-1.
* Have at least 1 measurable lesion according to RECIST 1.1 criteria.
* No prior treatment with abdominal radiotherapy, chemotherapy and PD-1/PD-L1 antibody.
* Adequate organs functions as defined by the following laboratory values (completed within 14 days prior to registration): (1) haemoglobin >= 90 g/L (no blood transfusion within 14 days)； (2) neutrophil count > 1.5x10^9/L； (3) platelet count >= 100x10^9/L； (4) total bilirubin <= 1.5xULN (upper limit of normal)； (5) blood glutamic transferase (ALT) or blood glutamic transferase (AST) <= 2.5xULN (6) endogenous creatinine clearance >= 60 ml/min (Cockcroft's AST). (ALT) or blood albumin transaminase (AST) <= 2.5xULN； (6) endogenous creatinine clearance >= 60 ml/min (Cockcroft-Gault formula)； (7) cardiac Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) >= 50%. (8) International normalised ratio (INR) of prothrombin time ≤ 1.5 and partial thromboplastin time (APTT) ≤ 1.5 times the upper limit of normal in patients who have not received anticoagulation. Patients receiving full or parenteral anticoagulant therapy may enter a clinical trial as long as the dose of anticoagulant has been stable for at least 2 weeks prior to entry into the clinical study and the results of coagulation assays are within the limits of local therapy.
* No congestive heart failure, unstable angina, unstable arrhythmia in the last 6 months.
* No previous severe haematopoietic, cardiac, pulmonary, hepatic or renal abnormalities or immunodeficiencies.
* Patient must be able to understand the potential risks and benefits associated with this study. Patient able to give informed consent and would likely to comply with the study parameters.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients with a history of other malignant diseases in the last 5 years, except cured skin cancer and cervical cancer in situ.
* Patients with a history of uncontrolled epilepsy, central nervous system disease or psychiatric disorders whose clinical severity, in the judgement of the investigator, may prevent the signing of informed consent or affect the patient's adherence to drug therapy.
* Severe heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) class II or worse congestive heart failure or severe arrhythmia requiring pharmacological intervention, or a history of myocardial infarction within the last 12 months.
* Organ transplants requiring immunosuppressive therapy
* Active infection or, in the investigator's judgement, significant haematological, renal, metabolic, gastrointestinal, endocrine function or metabolic disorders, or other serious uncontrolled concomitant disease
* Allergy to any of the study drug ingredients
* History of immunodeficiency, including HIV-positive or other acquired or congenital immunodeficiency diseases, or history of organ transplantation, or other immune-related diseases requiring long-term oral hormone therapy
* During acute or chronic tuberculosis infection (patients with a positive T-spot test and suspicious tuberculosis foci on chest radiographs).
* Other conditions considered by the investigator to be unsuitable for enrolment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-01-10 (Estimated); Study Completion 2027-01-10 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 36 months
  From the beginning of treatment, record the treatment-related toxic reactions that occur in patients.
Serious adverse events | 36 months
  From the start of treatment, record any severe adverse reactions that occur in the patient.
1-year overall survival | The 1-year overall survival rate of patients after receiving treatment
  Record the 1-year overall survival rate of patients after receiving treatment

SECONDARY OUTCOMES:
Objective response rate | 36 months
  The lesions were evaluated according to the RECIST1.1 standard, and the proportion of patients with the best treatment response of CR and PR after treatment to the total number of evaluable cases was calculated.
Disease control rate | 36 months
  The lesions were evaluated according to the RECIST1.1 standard, and the proportion of patients with optimal treatment response of CR, PR, and SD after treatment was calculated based on the total number of evaluable cases.
Overall survival | 36 months
  The time from the first day of enrollment to the occurrence of death due to any reason. Patients who are still alive at the time of analysis will use the date of their last contact as the deadline.
R0 resection rate | 36 months
  The tumor was completely removed during surgery, and the resection margin was negative under microscopic observation.
Progression free survival | 36 months
  The time between the start of treatment and the observation of disease progression or death for any reason. Patients who are still alive at the time of analysis will use the date of their last contact as the cutoff date.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT06345599/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT06345599/ICF_001.pdf